CLINICAL TRIAL: NCT03957577
Title: A Prospective, Epidemiological, Cohort Study to Assess the Aetiology of Acute Exacerbations of Chronic Obstructive Pulmonary Disease in Japan
Brief Title: Etiology of Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD) in Japan
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 208636
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Asthma-COPD overlap syndrome; Acute exacerbations of chronic obstructive pulmonary disease; Acute Exacerbation and Respiratory Infections in COPD-Japan; Chronic bronchitis; Chronic obstructive pulmonary disease; Exacerbation; Microbiome; Quantitative polymerase chain reaction (qPCR); 16S ribosomal Ribonucleic acid (16S rRNA); Metagenomic analysis; Sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Participants with COPD or Asthma-COPD overlap syndrome (ACOS)
  Interventions: Other: Prospective observational cohort study

INTERVENTIONS:
Other: Prospective observational cohort study — Prospective observational cohort study

SUMMARY:
The purpose of this prospective, epidemiological, cohort study is to evaluate the lung microbiome in stable-state chronic obstructive pulmonary disease (COPD) in Japanese participants

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able and willing to comply with the requirements of the protocol.
* Participant must be aged greater than or equal to (>=)40 years to to less than or equal to (<=)80 years at the time of signing the informed consent form (ICF).
* Participants must have a record of a clinical diagnosis of COPD, ACOS or CB.
* Participants must have moderate to severe airflow limitation based on spirometry: FEV1 percent predicted normal >=30 to <=80 percent (%) and post-bronchodilator FEV1/forced vital capacity (FVC) ratio <0.7.
* Participants must be symptomatic at Screening, defined as having a CAT score >=10.
* Participants must have a documented history of at least 1 LRTI treated with antibiotics and/or oral/systemic corticosteroids.
* Participants must be current or former tobacco (cigarette) smokers with a smoking history of >=10 pack-years.
* Participants may be male or female. For female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding. Women of non-childbearing potential can also participate. A woman of childbearing potential must have had a highly sensitive negative urine pregnancy test.
* Participants should be able to provide a spontaneous or induced sputum sample of >=0.2 grams (g) at the Screening Visit.

Exclusion Criteria:

* Participants with a diagnosed respiratory disorder other than COPD, ACOS or CB.
* Participants with a diagnosis of alpha-1 antitrypsin deficiency as the underlying cause of COPD.
* Participants who have received antibiotics within 1 month of Screening or have received antibiotics for more than 30 days within 90 days prior to Screening; Except for those who have received and are currently receiving long-term treatment with low-dose macrolide: erythromycin <=600 milligrams (mg) per (/) day or clarithromycin <=200 mg/day.
* Participants who have received systemic corticosteroids (oral/intravenous/intramuscular) for more than 14 consecutive days within 90 days prior to giving informed consent.
* Participants who are unable to use or to comply with daily completion of the eDiary.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll participants with a recorded clinical diagnosis of COPD, ACOS or chronic bronchitis (CB), who have airflow limitation indicative of COPD according to Global Initiative for Chronic Obstructive Lung Disease and a recent history of lower respiratory tract infection (LRTI).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with first evaluable moderate or severe AECOPD that have infectious or non-infectious etiology | Up to Month 12
Microbiome composition of sputum in stable-state COPD as measured by bacterial ribosomal ribonucleic acid (rRNA) sequencing | Baseline (Screening visit or Month 0)

SECONDARY OUTCOMES:
Number of all-cause moderate and severe AECOPD per participants | Up to Month 12
Microbiome composition of sputum in stable-state COPD as measured by bacterial rRNA sequencing | Baseline (Screening visit or Month 0)
Microbiome composition of sputum during participant's first evaluable moderate or severe AECOPD | Up to Month 12
Number of participants with first evaluable sputum samples that are positive for potentially pathogenic viruses (overall and by species) and bacteria in stable state COPD as measured by bacterial culture or quantitative polymerase chain reaction (qPCR) | Baseline (Screening visit or Month 0)
Number of participants with first evaluable sputum samples that are positive for potentially pathogenic viruses (overall and by species) and bacteria during moderate or severe AECOPD as measured by bacterial culture or qPCR | Baseline (Screening visit or Month 0)
Number of EXACT events per participant over the course of 12 months | Up to Month 12
  An EXACT event is defined as an increase in EXACT score more than or equal to 12 points for 2 days or more than or equal to 9 points for 3 days, above the participant's mean Baseline score. Severity is indicated by the worst (i.e., highest) EXACT total score during the course of the event.
Number of AECOPD events | Up to Month 12
Severity of AECOPD according to healthcare utilization | Up to Month 12
Severity of EXACT events according to EXACT total score | Up to Month 12
Duration of AECOPD | Up to Month 12
Duration of EXACT events | Up to Month 12
Mean change in CAT score between stable-state COPD and participants' first evaluable moderate or severe AECOPD | Baseline (Screening visit or Month 0) and up to Month 12
  The CAT is a 8-item, participant-completed instrument that covers symptoms such as cough, phlegm, chest tightness and breathlessness, and disease impacts including physical activity, confidence, sleep and energy. Participants will be asked to score each item on a scale ranging from 0 (no symptom or impact at all) to 5 (maximal symptom or impact).
Mean change in CAT score over the course of 1 year | Baseline (Screening visit or Month 0) and up to Month 12
  The CAT is a 8-item, participant-completed instrument that covers symptoms such as cough, phlegm, chest tightness and breathlessness, and disease impacts including physical activity, confidence, sleep and energy. Participants will be asked to score each item on a scale ranging from 0 (no symptom or impact at all) to 5 (maximal symptom or impact).
Mean change in EXACT score | Baseline(Screening visit or Month 0) and up to Month 12
  EXACT is a validated, self-administered, 14-item daily diary that assesses 11 respiratory symptoms and 3 additional symptoms, which together characterize COPD exacerbations. The EXACT total score will range from 0 to 100, with higher scores indicating a more severe condition.
Mean change in E-RS COPD total and subscale scores between stable-state COPD and participants' first evaluable moderate or severe AECOPD | Baseline (Screening visit or Month 0) and up to Month 12
  The E-RS: COPD comprises 11 of the 14 items of the parent EXACT that are specifically related to respiratory symptoms and will be completed using the eDiary. The RS-Total score is computed by taking the sum of the items comprising the instrument, with scores ranging from 0 to 40, with higher scores indicating more severe respiratory symptoms.
Mean change in E-RS: COPD total and subscale scores over the course of 1 year | Baseline (Screening visit or Month 0) and up to Month 12
  The E-RS: COPD comprises 11 of the 14 items of the parent EXACT that are specifically related to respiratory symptoms and will be completed using the eDiary. The RS-Total score is computed by taking the sum of the items comprising the instrument, with scores ranging from 0 to 40, with higher scores indicating more severe respiratory symptoms.
Mean change in Forced expiratory volume in 1 second (FEV1) between stable-state COPD, during participants' first evaluable moderate or severe AECOPD | Baseline (Screening visit or Month 0) and up to month 12
Mean rate of AECOPD related healthcare resource utilization per participant | Up to Month 12
Mean rate of non-AECOPD related healthcare resource utilization per participant | Up to Month 12
Annual rate of AECOPD related healthcare resource utilization per participant | Up to Month 12
Annual rate of non-AECOPD related healthcare resource utilization per participant | Up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: No